CLINICAL TRIAL: NCT06030089
Title: Plasma Dosage of Venetoclax in the Follow-up of Acute Myeloid Leukemias Ineligible for Intensive Chemotherapy in the First Line of Treatment and Treated With Azacitidine + Venetoclax. Pilot Study VENETACIBLE
Brief Title: Plasma Dosage of Venetoclax in the Fup of AML Patients Treated With Aza + Ven
Acronym: VENETACIBLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 23-AOIP-01
Record Dates: First submitted 2023-08-18; First posted 2023-09-08 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Acute Myeloid Leukemia
Keywords: acute myeloid leukemia; venetoclax; azacitidine
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AML patients ineligible for intensive chemotherapy and treated with azacitidine and venetoclax (Experimental): Newly diagnosed AML patients
  Interventions: Other: Pharmacokinetic sampling; Other: Vital status determination; Other: Toxicity assessments; Drug: Venetoclax and azacitidine combination

INTERVENTIONS:
Other: Pharmacokinetic sampling — 4 blood withdrawals ( before treatment, Day 5, Day 9 and relapse or 12 months after start of treatment) for the plasma dosage of VEN and inhibition of its Bcl-2
Other: Vital status determination — Survival situation 12 months after start of treament
Other: Toxicity assessments — Toxicity events
Drug: Venetoclax and azacitidine combination — Response to treatment

SUMMARY:
The study proposes to correlate the plasma dosage of VEN with the inhibition of its Bcl-2 target during the first treatment cycle. VEN will be measured sequentially during the first treatment cycle and assess inhibition of its target by measuring the level of phosphorylation of Bcl-2 serine 70. In parallel, BH3 profiling will be evaluated sequentially. All these analyses will be correlated with treatment toxicity, response rate and overall patient survival. This pilot study will highlight the inter-individual variability of this AZA + VEN combination, and enable to launch a national study via the national cooperative groups to validate the results and thus ultimately propose a personalized treatment for patients benefiting from this combination.

ELIGIBILITY:
Inclusion criteria :

* Patient with acute myeloid leukemia (AML) not eligible for intensive chemotherapy
* Patients aged 18 or over
* Patient treated with the combination azacitidine (AZA) + venetoclax (VEN)
* Patient having signed the study informed consent form
* Patient with social security coverage

Exclusion criteria :

* Patients receiving treatment inhibiting or inducing Cytochrome CYP3A4
* Presence of an active, uncontrolled infection
* Patient participating or having participated in a clinical drug trial in the month prior to inclusion.
* Vulnerable persons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-02-26 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2025-03-03 (Actual)

PRIMARY OUTCOMES:
Plasmatic dosage | Before treatment
  Correlation of VEN plasma levels with inhibition of its Bcl-2 target
Plasmatic dosage | At Day 5 of 1st round of chemotherapies
  Correlation of VEN plasma levels with inhibition of its Bcl-2 target
Plasmatic dosage | At Day 9 of 1st round of chemotherapies
  Correlation of VEN plasma levels with inhibition of its Bcl-2 target
Plasmatic dosage | At 12 months after start of treatment or at relapse whichever comes first
  Correlation of VEN plasma levels with inhibition of its Bcl-2 target

SECONDARY OUTCOMES:
Overall survival | 1 year
  Evaluate the overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Cluzeau, Principal Investigator — CHU of Nice
Locations (2):
- France (2):
  - Hopital la Conception, Marseille
  - CHU de Nice, Nice

IPD SHARING:
Plan to Share IPD: No